CLINICAL TRIAL: NCT01015092
Title: Predicted 10-year Coronary Heart Disease Risk in HIV and Implications for Clinical Management: the CREATE Study
Brief Title: Cardiovascular Risk Evaluation and Antiretrovirals in HIV
Acronym: CREATE1
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: Guy's and St Thomas' NHS Foundation Trust (Other)
Responsible Party: Dr Barry Stephen Peters, Kings College London
Other Study IDs: 05/Q0702/156
Record Dates: First submitted 2009-11-16; First posted 2009-11-17 (Estimated); Last update posted 2009-11-17 (Estimated); Status verified 2009-11

CONDITIONS: Cardiovascular Risk; HIV Infections
Keywords: HIV; Cardiovascular; Coronary hear disease; HAART; antiretroviral
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- unselected HIV outpatient attendees: All HIV patients attending for general HIV care at 2 London Hospitals

SUMMARY:
The purpose of the study is to determine the main factors contributing to predicted 10 year cardiovascular risk in an HIV infected cohort, and the role of anti-HIV drug use in altering this risk

ELIGIBILITY:
Inclusion Criteria:

* Serologically proven HIV infection
* Attending general HIV outpatient clinic

Exclusion Criteria:

* Attending a specialist outpatient clinic which might lead to recruitment bias

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All HIV outpatients patients attending two London Hospitals
Sampling Method: Probability Sample
Enrollment: 1024 (Actual)
Dates: Start 2005-06; Primary Completion 2006-09 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
10 year predicted cardiovascular risk | AT time of clinic attendence

SECONDARY OUTCOMES:
coronary heart disease risk | at time of clinic attendence

CONTACTS AND LOCATIONS:
Overall Officials: Barry S Peters, MB BS. MD, Principal Investigator — King's College London
Locations (1):
- Guys & ST Thomas' Foundation Hospitals, London, United Kingdom